CLINICAL TRIAL: NCT01276288
Title: Investigation of Pharmacodynamic and Pharmacokinetic Interactions Between 25 mg BI 10773 and 25 mg Hydrochlorothiazide or 5 mg Torasemide Under Steady State Conditions in Patients With Type 2 Diabetes Mellitus in an Open-label, Randomised, Cross-over Trial
Brief Title: Pharmacodynamics and Pharmacokinetics of Empagliflozin and Torasemide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.42; 2010-019624-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Hydrochlorothiazide; Torsemide

ARMS (5):
- Reference 1 (Active Comparator): administration of BI 10773 once daily for 5 days (20 patients)
  Interventions: Drug: BI 10773
- Reference 2 (Active Comparator): administration of hydrochlorothiazide (HTC) once daily for 4 days (10 patients)
  Interventions: Drug: hydrochlorothiazide
- Reference 3 (Active Comparator): administration of torasemide (TOR) once daily for 4 days (10 patients)
  Interventions: Drug: torasemide
- Test 1 (Experimental): administration of BI 10773 + HTC once daily for 5 days (10 patients)
  Interventions: Drug: hydrochlorothiazide; Drug: BI 10773
- Test 2 (Experimental): administration of BI 10773 + TOR once daily for 5 days (10 patients)
  Interventions: Drug: BI 10773; Drug: torasemide

INTERVENTIONS:
Drug: BI 10773 — multiple oral doses
  Arms: Test 2
Drug: hydrochlorothiazide — multiple oral doses
  Arms: Test 1
Drug: torasemide — multiple oral doses
  Arms: Reference 3
Drug: BI 10773 — multiple oral doses
  Arms: Reference 1
Drug: torasemide — multiple oral doses
  Arms: Test 2
Drug: BI 10773 — multiple oral doses
  Arms: Test 1
Drug: hydrochlorothiazide — multiple oral doses
  Arms: Reference 2

SUMMARY:
The primary objective of the study is to investigate the effect of BI 10773, hydrochlorothiazide and torasemide on changes in serum and urine electrolytes. Furthermore the pharmacodynamic and pharmacokinetic interactions between BI 10773 and diuretics should be assessed.

ELIGIBILITY:
Inclusion criteria:

1. male and female patients of type 2 diabetes

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.42.1 Boehringer Ingelheim Investigational Site, Neuss, Germany

REFERENCES:
- [Derived] Heise T, Jordan J, Wanner C, Heer M, Macha S, Mattheus M, Lund SS, Woerle HJ, Broedl UC. Pharmacodynamic Effects of Single and Multiple Doses of Empagliflozin in Patients With Type 2 Diabetes. Clin Ther. 2016 Oct;38(10):2265-2276. doi: 10.1016/j.clinthera.2016.09.001. Epub 2016 Sep 28. PMID 27692976
- [Derived] Heise T, Jordan J, Wanner C, Heer M, Macha S, Mattheus M, Lund SS, Woerle HJ, Broedl UC. Acute Pharmacodynamic Effects of Empagliflozin With and Without Diuretic Agents in Patients With Type 2 Diabetes Mellitus. Clin Ther. 2016 Oct;38(10):2248-2264.e5. doi: 10.1016/j.clinthera.2016.08.008. Epub 2016 Sep 22. PMID 27666126
- [Derived] Heise T, Mattheus M, Woerle HJ, Broedl UC, Macha S. Assessing pharmacokinetic interactions between the sodium glucose cotransporter 2 inhibitor empagliflozin and hydrochlorothiazide or torasemide in patients with type 2 diabetes mellitus: a randomized, open-label, crossover study. Clin Ther. 2015 Apr 1;37(4):793-803. doi: 10.1016/j.clinthera.2014.12.018. Epub 2015 Jan 28. PMID 25636696

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, open-label, 2- way cross-over study. All patients received empagliflozin (EMPA). After 7days washout period, half of patients received hydrochlorothiazide (HCT), other half torasemide (TOR) on its own or with EMPA. Then HCT or TOR and its combination with EMPA were administered first, followed by EMPA after 7 days washout.
Groups:
- Empa / Empa+HCT: Patients received 25mg empagliflozin (Empa) orally in a form of a film-coated tablet once daily following an overnight fast of at least 10 hours (h). Following a wash-out period of seven days, 25mg hydrochlorothiazide (HCT) in a form of a film-coated tablet was administered orally once daily in combination with 25mg Empa.
- Empa+HCT/ Empa: Patients received 25mg hydrochlorothiazide (HCT) in a form of a film-coated tablet orally once daily in combination with 25mg Empa. Following a wash-out period of seven days 25 mg Empa was administered in a form of a film-coated tablet orally once daily following an overnight fast of at least 10 hours (h).
- Empa/ Empa+ TOR: Patients received 25mg Empa in a form of a film-coated tablet orally once daily following an overnight fast of at least 10 hours (h). Following a wash-out period of seven days, 5 mg torasemide (TOR) in combination with 25mg Empa was administered.
- Empa+TOR/ Empa: Patients received 5mg torasemide (TOR) in combination with 25mg Empa. Following a wash-out period of seven days, 25 mg Empa was administered in a form of a film-coated tablet orally once daily following an overnight fast of at least 10 hours (h).
Period: Overall Study
Arm/Group | Empa / Empa+HCT | Empa+HCT/ Empa | Empa/ Empa+ TOR | Empa+TOR/ Empa
Started | 7 | 6 | 5 | 5
Received EMPA | 6 | 5 | 5 | 5
Received EMPA+HCT | 5 | 5 | 0 | 0
Received EMPA+TOR | 0 | 0 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) that includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Overall Patients: A randomised, open-label, multiple-dose, 2- way cross-over study. All patients received 25 mg empagliflozin in a form of a film-coated tablet orally once daily following an overnight fast of at least 10 hours (h) (days 1 to 5). Following a wash-out period of seven days, half of the patients received 25 mg hydrochlorothiazide (HCT) either on its own in a form of a film-coated tablet orally once daily (days 1 to 4) or in combination with 25 mg empagliflozin ( days 5 to 9), while the other half of the patients received 5 mg torasemide (TOR) either on its own (days 1 to 4) or in combination with the 25 mg empagliflozin ( days 5 to 9). This sequence was then reversed so that the HCT or TOR and its combination with 25 mg empagliflozin were administered first in a same manner as stated above, followed by 25 mg empagliflozin after seven days wash out period.
Arm/Group | Overall Patients
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Clearance of Sodium, Potassium, Creatinine, Magnesium, Chloride,Calcium, Phosphate and Uric Acid From Baseline
Description: Change in clearance of sodium, potassium, creatinine, magnesium, chloride,calcium, phosphate and uric acid from baseline, where baseline is defined as the value obtained from the last 24-h collection period before the first drug administration in the first treatment period.
  The mean change from baseline was evaluated as:
  Empa: day 5- baseline, HCT: day 4-baseline, TOR: day 4-baseline, Empa+ HCT: day 9- baseline, Empa+ TOR: day 9- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: 24 hour sampling interval at baseline and then day 5 for Empa, day 4 for TOR and HCT, day 9 for Empa+TOR and Empa+HCT
Population: Pharmacodynamic (PD) analysis set completers includes all evaluable patients of the treated set who provide a baseline and at least one on-treatment observation for at least one primary (PD) endpoint under any treatment without important protocol violations relevant to the evaluation of PD and who continued the trial as planned
Measure: Mean (Standard Error); unit: ml/min
Groups:
- Empagliflozin (Empa): Empagliflozin (Empa) 25 mg administered once daily for 5 days
- Hydrochlorothiazide (HCT): Hydrochlorothiazide (HCT) 25 mg administered once daily for 4 days
- Torasemide (TOR): Torasemide (TOR) 5 mg administered once daily for 4 days
- Empa+ HCT: Empagliflozin (Empa) 25 mg + Hydrochlorothiazide (HCT) 25 mg administered once daily for 5 days
- Empa + TOR: Empagliflozin (Empa) 25 mg + Torasemide (TOR) 5 mg administered once daily for 5 days
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
ml/min
  Sodium | -0.031 (0.038) | -0.055 (0.044) | -0.071 (0.083) | 0.143 (0.036) | -0.004 (0.088)
  Chloride | -0.129 (0.042) | -0.058 (0.056) | -0.157 (0.064) | 0.114 (0.044) | -0.117 (0.088)
  Potassium | 2.040 (0.492) | 2.205 (0.539) | -0.518 (0.585) | 4.125 (0.634) | 2.324 (0.832)
  Magnesium | 0.398 (0.171) | 1.826 (0.288) | 1.148 (0.206) | 1.115 (0.181) | 0.209 (0.227)
  Calcium | -0.326 (0.087) | -0.299 (0.094) | -0.065 (0.108) | -0.407 (0.102) | -0.174 (0.105)
  Phosphate | 5.275 (0.842) | 4.633 (1.342) | 4.368 (1.342) | 2.795 (1.382) | 2.359 (1.379)
  Uric Acid | 6.377 (1.100) | -0.476 (0.637) | -1.310 (0.924) | 5.065 (1.376) | 4.359 (1.533)
  Creatinine | 3.167 (4.306) | -7.034 (5.494) | -4.250 (6.574) | -10.126 (7.989) | -11.768 (7.135)

2. Primary Outcome: Change in Urinary Excretion in a 24-hour Period of Sodium, Potassium, Magnesium, Chloride, Calcium, Phosphate, Creatinine, Uric Acid, Glucose From Baseline
Description: Change in urinary excretion in a 24-hour period of sodium, potassium, magnesium, chloride, calcium, phosphate, creatinine, uric acid, glucose from baseline, where baseline was defined as the value obtained from the last 24-hour (h) collection period before the first drug administration in the first treatment period. This applies also to sodium excretion in urine, which is additionally obtained one day before the drug administration before the second period.
  The mean change from baseline was evaluated as:
  Empa: day 5- baseline, HCT: day 4-baseline, TOR: day 4-baseline, Empa+ HCT: day 9- baseline, Empa+ TOR: day 9- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: 24 hour sampling interval at baseline and then day 5 for Empa, day 4 for TOR and HCT, day 9 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mmol/day
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mmol/day
  Sodium | -4.300 (7.777) | -11.700 (8.495) | -13.700 (16.445) | 28.900 (7.512) | 1.200 (17.068)
  Chloride | -16.300 (6.363) | -12.300 (7.939) | -22.000 (9.421) | 11.400 (6.092) | -14.600 (12.120)
  Potassium | 10.370 (3.171) | 6.200 (3.008) | -6.990 (3.920) | 15.790 (2.963) | 8.460 (5.288)
  Magnesium | 1.190 (0.236) | 2.270 (0.387) | 1.720 (0.263) | 2.030 (0.225) | 1.050 (0.280)
  Calcium | -1.160 (0.281) | -1.020 (0.299) | -0.430 (0.377) | -1.360 (0.294) | -0.740 (0.306)
  Phosphate | 9.250 (1.198) | 9.000 (2.261) | 4.900 (1.900) | 8.300 (2.103) | 5.000 (2.357)
  Creatinine | 0.091 (0.043) | -0.078 (0.058) | -0.073 (0.045) | 0.022 (0.041) | -0.040 (0.068)
  Uric acid | 1.641 (0.334) | -0.037 (0.251) | -0.500 (0.349) | 1.555 (0.327) | 1.244 (0.493)
  Glucose | 599.449 (60.015) | 17.584 (8.161) | 17.932 (25.477) | 685.233 (68.035) | 740.910 (54.134)

3. Primary Outcome: Change in Urinary Excretion in a 24-hour Period of N-terminal Telopeptide (NTx) From Baseline
Description: Change in urinary excretion in a 24-hour period of N-terminal telopeptide (NTx) from baseline, where baseline was defined as the value obtained from the last 24-hour (h) collection period before the first drug administration in the first treatment period.
  The mean change from baseline was evaluated as:
  Empa: day 5- baseline, HCT: day 4-baseline, TOR: day 4-baseline, Empa+ HCT: day 9- baseline, Empa+ TOR: day 9- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: 24 hour sampling interval at baseline and then day 5 for Empa, day 4 for TOR and HCT, day 9 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: nM BCE/ mMC
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
nM BCE/ mMC | 6.010 (1.334) | 0.730 (2.704) | 2.030 (0.723) | 1.380 (3.429) | 3.900 (1.424)

4. Primary Outcome: Change in Serum Osmolality From Baseline
Description: Changes in serum osmolality from baseline based on a blood sample.
  Baseline was defined as the measurement obtained before the first drug administration in the first period.
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mOsm/Kg
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mOsm/Kg | 3.950 (3.748) | -7.500 (3.519) | -5.500 (2.915) | -2.200 (3.972) | 10.500 (3.625)

5. Primary Outcome: Change in Serum Concentration of Sodium, Potassium, Magnesium, Calcium, Chloride, Phosphate, Glucose and Urea From Baseline
Description: Change in serum concentration of sodium, potassium, magnesium, calcium, chloride, phosphate, glucose and urea from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mmol/L
  Sodium | 1.500 (0.447) | -0.500 (0.401) | 0.200 (0.573) | -0.100 (0.433) | 1.600 (1.222)
  Potassium | -0.170 (0.107) | -0.470 (0.087) | -0.200 (0.087) | -0.530 (0.091) | -0.360 (0.097)
  Magnesium | 0.139 (0.011) | 0.025 (0.014) | 0.059 (0.010) | 0.130 (0.014) | 0.145 (0.019)
  Chloride | 2.050 (0.592) | -2.600 (0.521) | 1.000 (0.775) | -3.200 (1.365) | 2.100 (1.650)
  Calcium | -0.055 (0.023) | -0.040 (0.034) | -0.080 (0.020) | -0.010 (0.031) | -0.060 (0.037)
  Phosphate | 0.045 (0.031) | 0.060 (0.031) | -0.060 (0.034) | 0.170 (0.040) | 0.050 (0.045)
  Urea | 0.710 (0.153) | 0.650 (0.149) | 0.318 (0.220) | 1.504 (0.161) | 2.122 (0.429)
  Glucose | -1.123 (0.250) | 0.849 (0.177) | 0.527 (0.290) | -0.033 (0.168) | -0.526 (0.389)

6. Primary Outcome: Change in Serum Concentration of Creatinine and Uric Acid From Baseline
Description: Change in serum concentration of Creatinine and Uric acid from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 5- baseline, HCT: day 4-baseline, TOR: day 4-baseline, Empa+ HCT: day 9- baseline, Empa+ TOR: day 9- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 5 for Empa, day 4 for TOR and HCT, day 9 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
umol/L
  Creatinine | 2.175 (1.585) | -0.340 (1.441) | -2.180 (1.811) | 6.280 (2.764) | 3.570 (2.348)
  Uric acid | -64.950 (24.763) | 24.200 (9.087) | -4.700 (9.164) | -31.000 (18.582) | -48.200 (12.984)

7. Primary Outcome: Change in Serum Concentration of Alkaline Phosphatase (ALP) From Baseline
Description: Change in serum concentration of ALP from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
U/L | 2.750 (0.878) | 3.000 (1.274) | 2.400 (0.859) | 6.500 (1.515) | 5.800 (1.788)

8. Primary Outcome: Change in Serum Concentration of Renin, Intact Parathyroid Hormone (iPTH) and 1,25-dihydroxyvitamin D From Baseline
Description: Change in serum concentration of Renin, intact parathyroid hormone (iPTH) and 1,25-dihydroxyvitamin D from baseline , where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
pg/mL
  Renin | -0.960 (4.155) | 16.150 (8.276) | 2.550 (1.882) | 32.760 (16.863) | 17.050 (3.645)
  iPTH | 8.265 (1.593) | 6.160 (1.880) | 6.910 (2.059) | 9.280 (1.619) | 12.190 (3.233)
  1,25-dihydroxyvitamin D | 0.230 (3.488) | 1.560 (4.029) | 3.530 (5.123) | -5.060 (4.070) | -0.970 (4.329)

9. Primary Outcome: Change in Serum Concentration of Aldosterone From Baseline
Description: Change in serum concentration of Aldosterone from baseline , where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
nmol/L | -0.018 (0.020) | 0.099 (0.056) | 0.023 (0.018) | 0.124 (0.068) | 0.123 (0.069)

10. Primary Outcome: Change in Serum Concentration of Fibroblast Growth Factor-23 (FGF- 23) From Baseline
Description: Change in serum concentration of fibroblast growth factor-23 (FGF- 23) from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline, The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: RU/mL
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
RU/mL | 50.305 (23.759) | 29.050 (25.952) | -0.680 (5.465) | 109.860 (53.745) | 13.820 (4.739)

11. Primary Outcome: Change in Urea Concentration in Urine
Description: Change in urea concentration in urine from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mmol/L | -1.515 (14.048) | 67.570 (29.271) | 35.710 (34.666) | 11.780 (9.819) | 48.690 (31.445)

12. Primary Outcome: Change in Urine pH From Baseline
Description: Change in urine pH from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: pH
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
pH | -0.132 (0.161) | -0.452 (0.291) | -0.147 (0.062) | -0.448 (0.259) | 0.130 (0.191)

13. Primary Outcome: Change in Urine Osmolality From Baseline
Description: Change in urine osmolality from baseline, where baseline was defined as the measurement obtained before first drug administration in the first period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mOsm/kg
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mOsm/kg | 223.15 (34.850) | -3.900 (43.239) | -5.800 (54.743) | 217.700 (31.430) | 330.400 (45.645)

14. Primary Outcome: Changes in Bicarbonate Concentrations of Calcium, Bicarbonate Ions and Base Excess in Capillary or Arterialised Blood From Baseline
Description: Changes in bicarbonate concentrations of calcium, bicarbonate ions and base excess in capillary or arterialised blood from baseline, where baseline was defined as the last measurement before trial drug administration of each treatment period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The means for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mmol/ L
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
mmol/ L
  Bicarbonate concentrations of calcium | -1.090 (0.309) | 2.020 (0.397) | -0.400 (0.450) | 1.860 (0.445) | -1.590 (0.580)
  bicarbonate ions | -0.049 (0.012) | -0.043 (0.023) | -0.041 (0.018) | -0.053 (0.015) | -0.049 (0.015)
  Base excess | -1.045 (0.284) | 1.640 (0.325) | -0.420 (0.386) | 1.720 (0.432) | -1.450 (0.576)

15. Primary Outcome: Change in pH in Capillary or Arterialised Blood From Baseline
Description: Change in pH in capillary or arterialised blood from baseline, where baseline was defined as the last measurement before trial drug administration of each treatment period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: pH
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
pH | -0.006 (0.004) | 0.003 (0.007) | -0.002 (0.006) | 0.008 (0.008) | -0.005 (0.008)

16. Primary Outcome: Change in Body Weight From Baseline
Description: Change in body weight from baseline , where baseline was defined as the last measurement before trial drug administration of each treatment period
  The mean change from baseline was evaluated as:
  Empa: day 6- baseline, HCT: day 5-baseline, TOR: day 5-baseline, Empa+ HCT: day 10- baseline, Empa+ TOR: day 10- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: baseline and then day 6 for Empa, day 5 for TOR and HCT, day 10 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: kg
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
kg | -1.365 (0.535) | -1.040 (0.227) | -0.380 (0.149) | -2.030 (0.344) | -1.750 (0.328)

17. Primary Outcome: Change in Urinary Weight From Baseline
Description: Change from baseline in urinary weight in a 24 hour (h)- collection period, where baseline is the last 24-h collection period before first trial drug administration in each treatment period.
  The mean change from baseline was evaluated as:
  Empa: day 5- baseline, HCT: day 4-baseline, TOR: day 4-baseline, Empa+ HCT: day 9- baseline, Empa+ TOR: day 9- baseline,
  The mean for the Empa arm represent combined adjusted means of all four sequences that is Empa administered before or after the administration of either TOR, HCT and their combination with Empa
Time Frame: 24 hour sampling interval at baseline and then day 5 for Empa, day 4 for TOR and HCT, day 9 for Empa+TOR and Empa+HCT
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: g/day
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 20 | 10 | 10 | 10 | 10
g/day | 134.700 (95.358) | -55.300 (67.517) | -39.000 (106.642) | 429.000 (92.357) | 353.200 (116.293)

18. Primary Outcome: The Change in Micturition Frequency From the Baseline
Description: For this endpoint the change in total micturition frequency from the baseline was only examined for EMPA where baseline was defined as the day before the first drug administration.
Time Frame: Baseline and day 5
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: voids per day
Arm/Group | Empagliflozin (Empa)
Number analyzed (Participants) | 20
voids per day | 1.600 (0.478)

19. Primary Outcome: The Change in Total Muscle Sympathetic Nerve Activity (MSNA) From Off- Treatment
Description: The change in total Muscle sympathetic nerve activity (MSNA) that represents an area under the curve of all C-fiber action potentials per minute. This endpoint was evaluated only for Empa. For this endpoint a baseline value was not defined. However, the parameters obtained at 2 measurements time points during the trial were compared.
Time Frame: One day before the drug administration, then day 4 after the first drug administration
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: action potentials per min
Arm/Group | Empagliflozin (Empa)
Number analyzed (Participants) | 20
action potentials per min | 0.241 (0.354)

20. Secondary Outcome: Area Under the Concentration-time Curve of Empa in Plasma (AUCτ,ss)
Description: Area under the concentration-time curve of Empa in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 post-dose on Day 5 with EMPA alone and on Day 9 with EMPA plus diuretic. The Pre-dose values were averaged over Days 1 to 4 with EMPA alone and on Days 7 & 8 with EMPA plus diuretic
Population: Pharmacokinetic (PK) set, including all patients of the treated set who provide at least one observation for at least one secondary PK endpoint of AUC τ,ss or C max,ss for any analyte under any treatment without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empagliflozin (Empa) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 21 | 10 | 10
nmol*h/L | 4990 (21.1) | 5570 (25.2) | 5260 (19.1)
Statistical Analysis 1: Comparison: Empagliflozin (Empa) vs Empa+ HCT; Only patients in sequences Empa/Empa+HCT were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0092, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa plus HCT divided by Empa; Model was adjusted for sequence, period and treatment as fixed effects while subjects within sequences as random effect; Geometric mean ratio = 107.08, 90% CI 2-sided [97.11 to 118.07], Standard Deviation 11.8 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 2: Comparison: Empagliflozin (Empa) vs Empa + TOR; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0030, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa plus TOR divided by Empa; Model was adjusted for sequence, period and treatment as fixed effects while subjects within sequences as random effect; Geometric mean ratio = 107.83, 90% CI 2-sided [100.14 to 116.11], Standard Deviation 8.9 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

21. Secondary Outcome: Maximum Measured Concentration of Empa in Plasma (Cmax, ss)
Description: Maximum measured concentration of Empa in plasma (Cmax, ss) at steady state
Time Frame: as for outcome 20
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin (Empa) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 21 | 10 | 10
nmol/L | 939 (21.4) | 1030 (31.2) | 949 (21.9)
Statistical Analysis 1: Comparison: Empagliflozin (Empa) vs Empa+ HCT; Only patients in sequences Empa/Empa+HCT were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0199, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ HCT divided by Empa; Model was adjusted for sequence, period and treatment as fixed effects while subjects within sequences as random effect; Geometric mean ratio = 102.78, 90% CI 2-sided [88.55 to 119.29], Standard Deviation 18.3 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 2: Comparison: Empagliflozin (Empa) vs Empa + TOR; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0086, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR divided by Empa; Model was adjusted for sequence, period and treatment as fixed effects while subjects within sequences as random effect; Geometric mean ratio = 107.50, 90% CI 2-sided [97.90 to 118.04], Standard Deviation 11.3 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

22. Secondary Outcome: Area Under the Concentration-time Curve of HCT in Plasma (AUCτ,ss)
Description: Area under the concentration-time curve of HCT in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 post-dose on Day 4 with HCT alone and on Day 9 with EMPA plus HCT. The Pre-dose values were averaged over Days 1 to 3 with HCT alone and on Days 7 & 8 with EMPA plus HCT
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- HCT+ Empa: Hydrochlorothiazide (HCT) 25 mg followed by Empagliflozin (Empa) 25 mg administered once daily for 5 days
Arm/Group | Hydrochlorothiazide (HCT) | HCT+ Empa
Number analyzed (Participants) | 11 | 10
ng*h/mL | 1040 (17.9) | 1000 (18.7)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCT) vs HCT+ Empa; Only patients in sequences Empa/Empa+HCT were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0008, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa plus HCT divided by HCT; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 96.27, 90% CI 2-sided [89.08 to 104.05], Standard Deviation 9.6 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

23. Secondary Outcome: Maximum Measured Concentration of HCT in Plasma (Cmax, ss)
Description: Maximum measured concentration of HCT in plasma (Cmax, ss) at steady state
Time Frame: as for outcome 22
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Hydrochlorothiazide (HCT) | HCT+ Empa
Number analyzed (Participants) | 11 | 10
ng/mL | 203 (31.5) | 205 (30.3)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCT) vs HCT+ Empa; Only patients in sequences Empa/Empa+HCT were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0114, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ HCT divided by HCT; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 101.77, 90% CI 2-sided [88.63 to 116.85], Standard Deviation 17.1 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

24. Secondary Outcome: Area Under the Concentration-time Curve of TOR in Plasma (AUCτ,ss)
Description: Area under the concentration-time curve of TOR in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 post-dose on Day 4 with TOR alone and on Day 9 with EMPA plus TOR. The Pre-dose values were averaged over Days 1 to 3 with TOR alone and on Days 7 & 8 with EMPA plus TOR
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- TOR+ Empa: Torasemide (TOR) 5 mg and Empagliflozin (Empa) 25 mg administered once daily for 5 days
- TOR Metabolite (TOR-M1): TOR metabolite with one-tenth of pharmacological activity of TOR after TOR undergoes extensive hepatic metabolism.
- TOR Metabolite (TOR-M3): TOR metabolite which pharmacological activity is equal to TOR after TOR undergoes extensive hepatic metabolism.
- TOR-M1+ Empa: TOR metabolite with one-tenth of pharmacological activity of TOR after TOR undergoes extensive hepatic metabolism in combination with Empa 25 mg
- TOR-M3 + Empa: TOR metabolite which pharmacological activity is equal to TOR after TOR undergoes extensive hepatic metabolism in combination with Empa 25 mg
Arm/Group | Torasemide (TOR) | TOR+ Empa | TOR Metabolite (TOR-M1) | TOR Metabolite (TOR-M3) | TOR-M1+ Empa | TOR-M3 + Empa
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng*h/mL | 1320 (14.0) | 1340 (16.1) | 74.8 (15.9) | 40.5 (23.9) | 78.1 (17.7) | 41.8 (18.2)
Statistical Analysis 1: Comparison: Torasemide (TOR) vs TOR+ Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p < 0.0001, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa plus TOR divided by TOR; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 101.44, 90% CI 2-sided [99.06 to 103.88], Standard Deviation 2.9 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 2: Comparison: TOR Metabolite (TOR-M1) vs TOR-M1+ Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p < 0.0001, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR-M1 divided by TOR-M1; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 104.42, 90% CI 2-sided [100.39 to 108.62], Standard Deviation 4.8 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 3: Comparison: TOR Metabolite (TOR-M3) vs TOR-M3 + Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0005, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR-M3 divided by TOR-M3; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 103.19, 90% CI 2-sided [95.93 to 111.01], Standard Deviation 8.9 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

25. Secondary Outcome: Maximum Measured Concentration of TOR in Plasma (Cmax, ss)
Description: Maximum measured concentration of Empa in plasma (Cmax, ss) at steady state
Time Frame: as for outcome 24
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Torasemide (TOR) | TOR+ Empa | TOR Metabolite (TOR-M1) | TOR Metabolite (TOR-M3) | TOR-M1+ Empa | TOR-M3 + Empa
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng/mL | 710 (19.1) | 741 (12.9) | 42.6 (23.0) | 8.58 (12.3) | 43.8 (18.0) | 8.79 (16.8)
Statistical Analysis 1: Comparison: Torasemide (TOR) vs TOR+ Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0066, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR divided by TOR; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 104.43, 90% CI 2-sided [93.81 to 116.25], Standard Deviation 13.1 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 2: Comparison: TOR Metabolite (TOR-M1) vs TOR-M1+ Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p = 0.0012, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR-M1 divided by TOR-M1; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 102.67, 90% CI 2-sided [94.13 to 111.97], Standard Deviation 10.6 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities
Statistical Analysis 3: Comparison: TOR Metabolite (TOR-M3) vs TOR-M3 + Empa; Only patients in sequences Empa/Empa+TOR were included; Test type: Non-Inferiority or Equivalence — No formal testing in a confirmatory sense; p < 0.0001, ANOVA — p-value for ratio outside interval 80-125% Ratio calculated as Empa+ TOR-M3 divided by TOR-M3; Model was adjusted for treatment as fixed effect and subject as random effect; Geometric mean ratio = 102.42, 90% CI 2-sided [97.65 to 107.42], Standard Deviation 5.8 — Standard deviation is actually the geometric coefficient of variation (gCV) reflecting intra-subject variabilities

26. Primary Outcome: Urinary Sodium Excretion Over 24-hour run-in Periods
Description: Urinary sodium excretion over 24-hour run-in periods to assess the harmonisation of electrolytes after intake of a standardised diet
Time Frame: Day 3, 2 and 1 before the first drug administration
Population: PD analysis set completers
Measure: Mean (Standard Error); unit: mmol/day
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR)
Number analyzed (Participants) | 20 | 10 | 10
mmol/day
  3 days before the drug administration | 198.50 (20.30) | 211.10 (9.37) | 217.90 (27.77)
  2 days before the drug administration | 174.35 (10.26) | 183.30 (13.15) | 178.70 (13.00)
  1 day before the drug administration | 163.90 (8.57) | 170.10 (7.58) | 179.10 (8.87)

27. Secondary Outcome: Number of Subjects With Clinical Relevant Abnormalities in Vital Signs, Clinical Laboratory Tests, 12-lead Resting Electrocardiogram (ECG), Physical Examination and Assessment of Tolerability by the Investigator
Description: Number of subjects with clinical relevant abnormalities in vital signs (blood pressure, pulse rate), 12-lead resting electrocardiogram (ECG), clinical laboratory tests (haematology, clinical chemistry, urinalysis, and monitoring of fasting plasma glucose), physical examination and assessment of tolerability by the investigator.
  New abnormal findings were reported as Adverse Events (AE). Only Alanine aminotransferase normal under system organ class investigations was determined as an existing AE.
Time Frame: From first drug administration until up to 14 days after the last drug administration, up to 35 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Number analyzed (Participants) | 21 | 11 | 10 | 10 | 10
participants | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until up to 14 days after the last drug administration, up to 35 days
Arm/Group | Empagliflozin (Empa) | Hydrochlorothiazide (HCT) | Torasemide (TOR) | Empa+ HCT | Empa + TOR
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/21 | 1/11 | 0/10 | 4/10 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin (Empa) (N=21) | Hydrochlorothiazide (HCT) (N=11) | Torasemide (TOR) (N=10) | Empa+ HCT (N=10) | Empa + TOR (N=10)
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 2 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.